CLINICAL TRIAL: NCT03738423
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study Investigating the Efficacy, Safety, and Pharmacokinetic Profiles of REGN3500 Administered to Adult Patients With Moderate-to- Severe Atopic Dermatitis
Brief Title: Efficacy, Safety, and Pharmacokinetic Profiles of REGN3500 Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3500-AD-1805; 2018-001544-64 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis
Keywords: Moderate; Severe
MeSH Terms: conditions — Dermatitis, Atopic; Lymphoma, Follicular | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment 1 (Experimental)
  Interventions: Drug: REGN3500; Drug: REGN3500-Matching Placebo
- Treatment 2 (Experimental)
  Interventions: Drug: REGN3500; Drug: REGN3500-Matching Placebo
- Treatment 3 (Experimental)
  Interventions: Drug: REGN3500; Drug: REGN3500-Matching Placebo
- Treatment 4 (Experimental)
  Interventions: Drug: REGN3500; Drug: REGN3500-Matching Placebo
- Treatment 5 (Experimental): Matching placebo
  Interventions: Drug: REGN3500-Matching Placebo

INTERVENTIONS:
Drug: REGN3500 — Administered subcutaneous (SC)
  Arms: Treatment 1; Treatment 2; Treatment 3; Treatment 4
Drug: REGN3500-Matching Placebo — Administered subcutaneous (SC)

SUMMARY:
The primary objective of the study is to assess the efficacy of REGN3500 monotherapy in Atopic dermatitis (AD), as well as understand the dose-response relationship, compared with placebo treatment, in adult patients with moderate-to-severe AD.

Secondary objectives are to:

* Assess the safety and tolerability of subcutaneous (SC) doses of REGN3500 monotherapy in adult patients with moderate-to-severe AD
* Assess the Pharmacokinetics (PK) of REGN3500 in adult patients with moderate-to-severe AD
* Assess the immunogenicity of REGN3500 in adult patients with moderate-to-severe AD

ELIGIBILITY:
Key Inclusion Criteria:

1. Chronic AD, according to American Academy of Dermatology Consensus Criteria (Eichenfield, 2014), that has been present for at least 3 years before the screening visit
2. Eczema Area and Severity Index (EASI) score ≥16 at the screening and baseline visits
3. IGA score ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at screening and baseline visits
4. ≥10% Body surface area (BSA) of AD involvement at the screening and baseline visits
5. Documented recent history (within 6 months before the screening visit) of inadequate response to topical AD medication(s) or for whom topical treatments are medically inadvisable

Key Exclusion Criteria:

1. Participation in a prior anti-Interleukin (IL)-33 medication clinical study
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
3. Having used any of the following treatments within 4 weeks before the baseline visit or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment:

   1. Immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, Interferon-gamma (IFN-γ), Janus kinase inhibitors, azathioprine, methotrexate, etc)
   2. Phototherapy for AD
4. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the baseline visit
5. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit
6. Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit
7. Known or suspected history of immunosuppression
8. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
9. Positive with hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (HCV Ab) at the screening visit
10. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Note: Other protocol defined Inclusion/Exclusion Criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (75):
- United States (27):
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Scottsdale, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, Little Rock, Arkansas
  - Regeneron Study Site, Fountain Valley, California
  - Regeneron Study Site, Fremont, California
  - Regeneron Study Site, Oceanside, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Jacksonville, Florida
  - Regeneron Study Site, Macon, Georgia
  - Regeneron Study Site, Skokie, Illinois
  - Regeneron Study Site, Evansville, Indiana
  - Regeneron Study Site, Overland Park, Kansas
  - Regeneron Study Site, Louisville, Kentucky
  - Regeneron Study Site, Saint Joseph, Michigan
  - Regeneron Study Site, Minneapolis, Minnesota
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Lebanon, New Hampshire
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Norman, Oklahoma
  - Regeneron Study Site, North Charleston, South Carolina
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Norfolk, Virginia
- Australia (2):
  - Regeneron Study Site, Kogarah
  - Regeneron Study Site, Melbourne
- Canada (5):
  - Regeneron Study Site, Calgary, Alberta
  - Regeneron Study Site, Hamilton, Ontario
  - Regeneron Study Site, Toronto, Ontario
  - Regeneron Study Site, Windsor, Ontario
  - Regeneron Study Site, Verdun, Quebec
- Czechia (4):
  - Regeneron Study Site, Brno
  - Regeneron Study Site, Náchod
  - Regeneron Study Site, Ostrava
  - Regeneron Study Site, Prague
- Germany (12):
  - Regeneron Study Site, Bad Bentheim
  - Regeneron Study Site, Berlin
  - Regeneron Study Site, Frankfurt
  - Regeneron Study Site, Hamburg
  - Regeneron Study Site, Hanau
  - Regeneron Study Site, Ibbenbueren
  - Regeneron Study Site, Leipzig
  - Regeneron Study Site, Lübeck
  - Regeneron Study Site, München
  - Regeneron Study Site, Münster
  - Regeneron Study Site, Tübingen
  - Regeneron Study Site, Witten
- Hungary (3):
  - Regeneron Study Site, Orosháza, Bekes County
  - Regeneron Study Site, Debrecen, Hajdú-Bihar
  - Regeneron Study Site, Budapest
- Japan (7):
  - Regeneron Study Site, Chūō
  - Regeneron Study Site, Hiroshima
  - Regeneron Study Site, Kanagawa
  - Regeneron Study Site, Kyoto
  - Regeneron Study Site, Shizuoka
  - Regeneron Study Site, Wakayama
  - Regeneron Study Site, Yamanashi
- Poland (5):
  - Regeneron Study Site, Krakow
  - Regeneron Study Site, Lodz
  - Regeneron Study Site, Szczecin
  - Regeneron Study Site, Warsaw
  - Regeneron Study Site, Wroclaw
- South Korea (5):
  - Regeneron Study Site, Bucheon-si
  - Regeneron Study Site, Busan
  - Regeneron Study Site, Gyeonggi-do
  - Regeneron Study Site, Incheon
  - Regeneron Study Site, Seoul
- Spain (4):
  - Regeneron Study Site, Barakaldo
  - Regeneron Study Site, Córdoba
  - Regeneron Study Site, Madrid
  - Regeneron Study Site, Santiago de Compostela
- Regeneron Study Site, Sheffield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 238 participants were screened at centers in North America (United States of America and Canada), Europe (Czech Republic, Germany, Hungary, Spain, and Poland), and Asia Pacific (Republic of Korea, Japan, and Australia). Out of which, 129 participants were randomized in this study.
Pre-assignment Details: Participants were randomized in 1:1:1:1:1 ratio to 1 of the 5 treatment groups: Placebo every 2 weeks (Q2W); REGN3500 30 milligrams (mg) every 8 weeks (Q8W); REGN3500 100 mg every 4 weeks (Q4W); REGN3500 300 mg Q4W and REGN3500 300 mg Q2W.
Groups:
- Placebo Q2W: Participants received 3 subcutaneous (SC) injections of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 4, 6, 10, 12, and 14.
- REGN3500 30 mg Q8W: Participants received 1 SC injection of REGN3500 (30 mg total dose) along with 2 SC injections of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 4, 6, 10, 12, and 14.
- REGN3500 100 mg Q4W: Participants received 1 SC injection of REGN3500 (100 mg total dose) along with 2 SC injections of placebo matched to REGN3500 on Day 1 and Week 8 and 1 SC injection of REGN3500 (100 mg total dose) in combination with 1 SC injection of placebo matched to REGN3500 at Weeks 4 and 12 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 6, 10, and 14.
- REGN3500 300 mg Q4W: Participants received 2 SC injections of REGN3500 (300 mg total dose) along with 1 SC injection of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of REGN3500 (300 mg total dose) at Weeks 4 and 12 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 6, 10, and 14.
- REGN3500 300 mg Q2W: Participants received 2 SC injections of REGN3500 (300 mg total dose) along with 1 SC injection of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of REGN3500 (300 mg total dose) at Weeks 2, 4, 6, 10, 12 and 14.
Period: Overall Study
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Started | 25 | 26 | 27 | 25 | 26
Treated | 25 | 26 | 26 | 24 | 26
Completed | 11 | 13 | 14 | 10 | 11
Not Completed | 14 | 13 | 13 | 15 | 15
Not completed — Withdrawal by Subject | 9 | 12 | 9 | 12 | 10
Not completed — Lack of Efficacy | 3 | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Randomized but never treated | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants and was based on the treatment allocated (as randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W | Total
Number analyzed (Participants) | 25 | 26 | 27 | 25 | 26 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (14.22) | 36.0 (16.41) | 37.0 (14.48) | 35.6 (12.56) | 38.8 (15.44) | 36.8 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 12 | 14 | 15 | 68
  Male | 11 | 13 | 15 | 11 | 11 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 0 | 0 | 7
  Not Hispanic or Latino | 24 | 24 | 22 | 25 | 23 | 118
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 8 | 5 | 11 | 10 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 3 | 2 | 14
  White | 13 | 14 | 20 | 11 | 14 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Scores on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. FAS included all randomized participants and was based on the treatment allocated (as randomized). Population: Here, "Number Analyzed" signifies those participants who were evaluable for this baseline characteristic.
  Scores on a scale
    number analyzed (Participants) | 25 | 26 | 27 | 24 | 26 | 128
    (all) | 30.3 (11.88) | 29.8 (12.00) | 33.6 (11.01) | 27.7 (10.68) | 32.7 (15.13) | 30.9 (12.25)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percent change from baseline in EASI score at Week 16 was reported. Values after first rescue treatment were set to missing.
Time Frame: Week 16
Population: FAS included all randomized participants and was based on the treatment allocated (as randomized). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
  Due to premature discontinuation, all statistical analyses were descriptive, and no hypothesis testing was performed.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Percentage of change | -33.5 (41.81) | -57.9 (31.65) | -52.7 (46.64) | -80.0 (10.54) | -54.0 (36.80)

2. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percent change from baseline in EASI score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of change | -18.9 (52.01) | -46.0 (45.35) | -48.7 (44.66) | -67.0 (28.74) | -56.1 (35.32)

3. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-50 (EASI-50) (Greater Than or Equal to [≥] 50 Percent [%] Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-50 (≥50% Improvement from baseline) at Week 16 were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Percentage of participants | 30.0 | 71.4 | 71.4 | 100 | 55.6

4. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-50 (EASI-50) (Greater Than or Equal to [≥] 50% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-50 (≥50% Improvement from baseline) at Week 16 were based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of participants | 25.0 | 60.0 | 62.5 | 77.8 | 60.0

5. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-75 (≥75% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Percentage of participants | 20.0 | 28.6 | 28.6 | 71.4 | 44.4

6. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-75 (≥75% Improvement from baseline) at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of participants | 16.7 | 30.0 | 25.0 | 55.6 | 40.0

7. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-90 (≥90% Improvement from baseline) at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Percentage of participants | 10.0 | 14.3 | 28.6 | 28.6 | 33.3

8. Secondary Outcome: Percentage of Participants Who Achieved Eczema Area and Severity Index-90 (EASI-90) (≥90% Improvement From Baseline) Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Percentage of participants who achieved EASI-90 (≥90% Improvement from baseline) at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of participants | 8.3 | 20.0 | 25.0 | 22.2 | 30.0

9. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Absolute change from baseline in EASI score at Week 16 based on observed values set to missing after rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Score on a scale | -7.8 (10.225) | -14.64 (8.489) | -14.81 (12.614) | -18.19 (6.298) | -13.79 (9.534)

10. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Absolute change from baseline in EASI score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Score on a scale | -4.10 (13.079) | -12.07 (11.764) | -13.83 (12.000) | -15.15 (8.299) | -14.68 (9.410)

11. Secondary Outcome: Percentage of Participants With Both Investigator Global Assessment (IGA) Score 0 or 1 (on 0 to 5 IGA Scale) and a Reduction From Baseline of ≥2 Points Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5 point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with both IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing IGA score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 10 | 7 | 7 | 7 | 9
Percentage of participants | 10.0 | 0.0 | 28.6 | 42.9 | 33.3

12. Secondary Outcome: Percentage of Participants With Both IGA Score 0 or 1 (on the 0 to 5 IGA Scale) and a Reduction From Baseline of ≥2 Points Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5 point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Participants with both IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of participants | 8.3 | 0.0 | 25.0 | 33.3 | 30.0

13. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Daily Peak Pruritus Numerical Rating Scale (NRS) Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Absolute change from baseline in weekly average of daily Peak Pruritus NRS score at Week 16 based on observed values set to missing after rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 8
Score on a scale | -0.53 (1.583) | -2.95 (3.791) | -4.22 (2.372) | -3.34 (2.628) | -3.12 (3.896)

14. Secondary Outcome: Absolute Change From Baseline in Weekly Average of Daily Peak Pruritus NRS Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Absolute Change From Baseline in Weekly Average of Daily Peak Pruritus NRS Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 8
Score on a scale | -0.51 (1.430) | -2.56 (3.563) | -4.19 (2.198) | -2.69 (2.799) | -3.12 (3.896)

15. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily Peak Pruritus NRS Score Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percent change from baseline in weekly average of daily peak pruritus NRS score at Week 16 based on observed values set to missing after rescue treatment was reported. Values after first rescue treatment were set to missing and participants with missing NRS score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 8
Percentage of change | -6.1 (20.65) | -31.6 (39.01) | -53.1 (29.65) | -43.1 (36.42) | -32.2 (47.46)

16. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily Peak Pruritus NRS Score Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percent change from baseline in weekly average of daily peak pruritus NRS score at Week 16 based on all observed values regardless of rescue treatment was reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 8
Percentage of change | -5.9 (18.62) | -27.5 (39.24) | -52.8 (27.47) | -33.9 (38.71) | -32.2 (47.46)

17. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) in Weekly Average of Peak Daily Pruritus NRS Score ≥4 Based on Observed Values Set to Missing After Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percentage of participants with improvement of weekly average of daily peak pruritus NRS score ≥4 from baseline to Week 16 based on observed values set to missing after rescue treatment were reported. Values after first rescue treatment were set to missing and participants with missing NRS score at Week 16 were counted as non-responders.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 8
Percentage of participants | 0.0 | 42.9 | 57.1 | 28.6 | 50.0

18. Secondary Outcome: Percentage of Participants With Improvement (Reduction From Baseline) in Weekly Average of Daily Peak Pruritus NRS Score ≥4 Based on All Observed Values Regardless of Rescue Treatment at Week 16
Description: Pruritus NRS was an assessment tool used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, using an electronic questionnaire (e-diary). Participants were asked the following question: how would you rate your itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Percentage of participants with improvement of weekly average of daily peak pruritus NRS score ≥4 from baseline to Week 16 based on all observed values regardless of rescue treatment were reported.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 11 | 10 | 8 | 9 | 8
Percentage of participants | 0.0 | 40.0 | 62.5 | 22.2 | 50.0

19. Secondary Outcome: Time to Onset of Effect on Pruritus (≥4-point Reduction of Weekly Average of Daily Peak Pruritus NRS From Baseline)
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?"
Time Frame: Week 16
Population: Time to event analysis performed for participants in FAS with baseline weekly peak NRS score ≥4 and at least one post-baseline weekly peak NRS score reduced ≥4 points from baseline. Time to event was calculated in weeks as the (date of first event - the date of first dose)/7. The event of NRS reduction ≥4 was based on observed data regardless of rescue use. Here 'n' = number of evaluable participants analyzed at specified time frame.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 5 | 6 | 8 | 6 | 4
Weeks | 6.6 (3.71) | 7.1 (4.74) | 7.1 (5.02) | 6.0 (4.29) | 5.8 (3.50)

20. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis (AD). Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Week 16
Population: FAS; All observed values, regardless of rescue treatment use; Here 'n' = number of evaluable participants at the specific timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of change | -12.7 (25.41) | -31.4 (22.67) | -39.2 (38.39) | -42.40 (20.00) | -40.5 (29.00)

21. Secondary Outcome: Absolute Change From Baseline in Percent Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement at Week 16
Description: BSA affected by AD will be assessed for each section of the body using the rule of nines (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined. The proportion assigned to different body regions is different in younger children as compared to older children (head and neck area is assigned a higher proportion in younger children as compared to older children).
Time Frame: Week 16
Population: FAS; All observed values regardless of rescue treatment use; Here 'n' = number of evaluable participants at the specific timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 12 | 10 | 8 | 9 | 10
Percentage of change | -2.74 (17.854) | -15.19 (16.509) | -11.43 (22.022) | -22.16 (15.783) | -20.99 (16.161)

22. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) up to Week 16
Description: Adverse Event (AE): any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. Serious AE (SAE): any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAE: AEs starting/worsening after first intake of study drug. TEAEs included: serious TEAEs and Non-serious TEAEs. AESI included: Anaphylactic or acute allergic reactions; Severe injection site reactions; Mycosis fungoides/other forms of cutaneous T-cell lymphoma; severe infections; any clinical endoparasitosis; Conjunctivitis, keratitis, or blepharitis; significant Alanine aminotransferase (ALT) elevation. Number of participants with TEAEs, Serious TEAES and AESIs from baseline up to Week 16 were reported.
Time Frame: Up to week 16
Population: The safety analysis set (SAF) included all randomized participants who received any study drug and was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 25 | 26 | 26 | 24 | 26
Participants
  Participants with TEAEs | 9 | 13 | 12 | 9 | 15
  Participants with Serious TEAEs | 0 | 0 | 0 | 0 | 2
  Participants with AESIs | 0 | 0 | 1 | 0 | 0

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESIs) up to Week 36
Description: AE: any untoward medical occurrence in a participant administered a study drug which may/may not have a causal relationship with study drug. SAE: any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAE: AEs starting/worsening after first intake of study drug. TEAEs included both Serious TEAEs and Non-serious TEAEs. AESI included: Anaphylactic or acute allergic reactions; Severe injection site reactions; Mycosis fungoides/other forms of cutaneous T-cell lymphoma; severe infections; any clinical endoparasitosis; Conjunctivitis, keratitis, or blepharitis; significant Alanine aminotransferase (ALT) elevation. Number of participants with TEAEs, Serious TEAES and AESIs from baseline up to Week 36 were reported.
Time Frame: Up to week 36
Population: SAF included all randomized participants who received any study drug and was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 25 | 26 | 26 | 24 | 26
Participants
  Participants with TEAEs | 11 | 14 | 14 | 13 | 15
  Participants with Serious TEAEs | 0 | 0 | 0 | 1 | 2
  Participants with AESIs | 0 | 0 | 1 | 0 | 0

24. Secondary Outcome: Serum Concentration of Functional REGN3500
Description: Serum Concentration of Functional REGN3500 was reported.
Time Frame: Baseline (Week 0), Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32 and 36
Population: The Pharmacokinetic (PK) analysis set included all randomized participants who received any study drug and who had at least 1 non-missing study drug concentration result following the first dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable at given time points.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 0 | 26 | 26 | 24 | 26
Milligrams per Liter (mg/L)
  Baseline (Week 0) |  | NA (NA) — Data were below the level of quantitation | 0.157 (0.800) | NA (NA) — Data were below the level of quantitation | NA (NA) — Data were below the level of quantitation
  Week 2: number analyzed (Participants) | 0 | 25 | 25 | 22 | 25
  Week 2 |  | 3.29 (2.70) | 7.35 (5.65) | 21.4 (9.83) | 22.0 (11.0)
  Week 4: number analyzed (Participants) | 0 | 22 | 21 | 23 | 21
  Week 4 |  | 2.33 (1.82) | 5.14 (3.73) | 14.3 (7.05) | 37.9 (15.2)
  Week 8: number analyzed (Participants) | 0 | 19 | 20 | 22 | 15
  Week 8 |  | 1.41 (1.99) | 9.27 (5.33) | 23.3 (10.4) | 51.4 (20.7)
  Week 12: number analyzed (Participants) | 0 | 14 | 14 | 17 | 13
  Week 12 |  | 2.63 (2.20) | 8.74 (6.37) | 30.3 (12.0) | 57.7 (26.3)
  Week 16: number analyzed (Participants) | 0 | 11 | 11 | 12 | 13
  Week 16 |  | 1.05 (0.733) | 10.6 (4.91) | 35.2 (17.3) | 60.8 (33.3)
  Week 20: number analyzed (Participants) | 0 | 13 | 8 | 9 | 9
  Week 20 |  | 0.523 (0.441) | 5.03 (3.93) | 12.4 (6.58) | 29.8 (23.5)
  Week 24: number analyzed (Participants) | 0 | 8 | 6 | 8 | 7
  Week 24 |  | 0.170 (0.157) | 2.23 (1.24) | 7.14 (5.22) | 12.1 (14.4)
  Week 28: number analyzed (Participants) | 0 | 8 | 6 | 6 | 7
  Week 28 |  | 0.0838 (0.109) | 1.08 (0.813) | 3.49 (2.76) | 6.70 (7.64)
  Week 32: number analyzed (Participants) | 0 | 8 | 6 | 6 | 8
  Week 32 |  | 0.0171 (0.0484) | 0.625 (0.560) | 1.93 (1.37) | 3.73 (5.41)
  Week 36: number analyzed (Participants) | 0 | 8 | 6 | 6 | 7
  Week 36 |  | NA (NA) — Data were below the level of quantitation | 0.299 (0.250) | 0.960 (0.741) | 1.02 (1.31)

25. Secondary Outcome: Number of Participants With Positive Treatment-Emergent Anti-REGN3500 Antibodies (ADA)
Description: Treatment-Emergent (TE) ADA was defined as any positive post baseline assay response when baseline results were negative or missing. Treatment-Emergent ADA responses were further classified as: - persistent (treatment-emergent positive ADA response detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period [based on nominal sampling time], with no ADA-negative samples in-between, regardless of any missing samples or a positive response at the last ADA sampling time point),- indeterminate (a positive assay response at the last collection time point only, regardless of any missing samples), - transient (not persistent/indeterminate, regardless of any missing samples). Number of participants with positive treatment-emergent anti-REGN3500 antibodies (ADA) were reported. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this endpoint.
Time Frame: Up to week 36
Population: The Anti-drug Antibodies (ADA) analysis set included all treated participants who received any amount of study drug (active or placebo [safety analysis set]) and had at least one non-missing anti-REGN3500 result following the first dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | REGN3500 30 mg Q8W | REGN3500 100 mg Q4W | REGN3500 300 mg Q4W | REGN3500 300 mg Q2W
Number analyzed (Participants) | 24 | 25 | 25 | 22 | 24
Participants
  TE Persistent | 0 | 0 | 0 | 0 | 0
  TE Transient | 0 | 0 | 0 | 0 | 0
  TE Indeterminate | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the end of study (Week 36) regardless of seriousness or relationship to investigational product (IP).
Groups:
- R3500 30 mg Q8W: Participants received 1 SC injection of REGN3500 (30 mg total dose) along with 2 SC injections of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 4, 6, 10, 12, and 14.
- R3500 100 mg Q4W; R3500 300 mg Q4W: Participants received 2 SC injections of REGN3500 (300 mg total dose) along with 1 SC injection of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of REGN3500 (300 mg total dose) at Weeks 4 and 12 and 2 SC injections of placebo matched to REGN3500 at Weeks 2, 6, 10, and 14.
- R3500 300 mg Q2W: Participants received 2 SC injections of REGN3500 (300 mg total dose) along with 1 SC injection of placebo matched to REGN3500 on Day 1 and Week 8 and 2 SC injections of REGN3500 (300 mg total dose) at Weeks 2, 4, 6, 10, 12 and 14.
Arm/Group | Placebo Q2W | R3500 30 mg Q8W | R3500 100 mg Q4W | R3500 300 mg Q4W | R3500 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 1/24 | 2/26
Other Adverse Events (participants affected / at risk) | 7/25 | 11/26 | 9/26 | 8/24 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=25) | R3500 30 mg Q8W (N=26) | R3500 100 mg Q4W (N=26) | R3500 300 mg Q4W (N=24) | R3500 300 mg Q2W (N=26)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=25) | R3500 30 mg Q8W (N=26) | R3500 100 mg Q4W (N=26) | R3500 300 mg Q4W (N=24) | R3500 300 mg Q2W (N=26)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9) | 5 (5) | 5 (5) | 6 (7)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The decision was made by the sponsor to terminate the study on 12 Feb 2020 due to lack of efficacy. Study enrollment was not complete at that time, therefore planned sample sizes were not met. Participants discontinued study drug and transitioned into the post-treatment follow-up period. As a result of the decision to terminate the study, all statistical analyses were descriptive and no hypothesis testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03738423/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03738423/SAP_001.pdf